CLINICAL TRIAL: NCT00490009
Title: Phase 2 Study of Bexxar in Relapsed/Refractory Diffuse Large Cell Lymphoma (DLCL)
Brief Title: Phase 2 Study of Bexxar in Relapsed/Refractory DLCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Susan Knox (Other)
Collaborators: Corixa Corporation (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Susan Knox, Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-10275; LYMNHL0019 (Other: OnCore); 30978 (Other: Stanford SPO)
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — tositumomab I-131; Acetaminophen; Diphenhydramine; Potassium Iodide; Lugol's solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bexxar + Total Body Irradiation (TBI) (Experimental): Bexxar will be administered with pre-medications acetaminophen, diphenhydramine, and potassium iodide (KI).
  Interventions: Drug: Bexxar; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Potassium Iodide (KI)

INTERVENTIONS:
Drug: Bexxar — Bexxar is a radioimmunotherapeutic drug, an antibody that specifically attaches to the CD20 antigen, which is present on the surfaces of B cells and B cell lymphoma cells. The radioactive isotope then gives off radiation, which kills the cells.
  Bexxar will be administered to provide the following patient-specific radiotherapy:
  * Platelet count of 150,000/mm³ = 75 cGy
  * Platelet count ≥ 100,000/mm³ but < 150,000/mm³ = 65 cGy
  Other Names: Tositumomab; iodine-131 tositumomab; I-131 tositumomab
Drug: Acetaminophen — As premedication 30 to 60 minutes before antibody infusion; 650 mg, oral. Used to as to relieve pain
  Other Names: Tylenol
Drug: Diphenhydramine — As premedication 30 to 60 minutes before antibody infusion; 50 mg, oral. Used to prevent inflammation or allergic reactions
  Other Names: Benadryl
Drug: Potassium Iodide (KI) — Administered to prevent thyroid blockage 130 mg orally 3 times a day,
  Other Names: Saturated solution potassium iodine (SSKI); Lugol's solution

SUMMARY:
The purpose of this study is to obtain safety and efficacy data using Bexxar in patients with relapsed/refractory diffuse large cell Non-Hodgkin's lymphoma (DLCL).

DETAILED DESCRIPTION:
There is a lack of efficacious treatment options for patients with relapsed/refractory diffuse large cell Non-Hodgkin's lymphoma (DLCL) who are not appropriate candidates for stem cell transplantation. DLCL is a relatively radiosensitive disease and patients with DLCL have been reported to respond to anti-CD20 monoclonal antibody (MAB) therapy. Therefore, radioimmunotherapy targeting CD20 is a rational and promising therapeutic approach for this patient population.

This study evaluated if Bexxar is safe and efficacious for diffuse large cell Non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed, diffuse large cell lymphoma (DLCL), CD20+ B-cell non-Hodgkin lymphoma (NHL) who have relapsed after chemotherapy or are chemotherapy resistant, without prior history of low grade NHL. The patient must have failed at least one chemotherapy regimen containing an anthracycline or equivalent chemotherapeutic agent.
* No anticancer treatment for three weeks prior to the treatment dose of Bexxar (6 weeks if Rituximab, nitrosourea or Mitomycin C)
* Fully recovered from all toxicities associated with prior surgery, radiation, chemotherapy or immunotherapy
* An Institutional Review Board (IRB)-approved signed informed consent
* Age 19 years or older
* Prestudy Karnofsky Performance Status of ≥ 70%
* Absolute neutrophil count (ANC) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hct > 30%
* Hgb > 9.0 gm%
* Bilirubin ≤ 2.0
* Creatinine ≤ 2.0
* Bone marrow involvement with lymphoma less than 25% (bilateral bone marrow) within 6 weeks of enrollment
* Acceptable birth control method for men and women
* Female patients who are not pregnant
* Not lactating

Exclusion Criteria:

* Prior myeloablative therapies with bone marrow transplantation or peripheral stem cell rescue
* Platelet count < 100,000/mm³
* Hypocellular bone marrow (≤ 15% cellularity)
* Marked reduction in bone marrow precursors of one or more cell lines
* History of failed stem cell collection
* Prior treatment with Fludarabine
* Prior radioimmunotherapy
* Presence of central nervous system (CNS) lymphoma
* Patients with known HIV or AIDS-related lymphoma
* Patients with evidence of myelodysplasia on bone marrow biopsy
* Patients who have received prior external beam radiation therapy to more than 25% of active bone marrow
* Patients who have received filgrastim or sargramostim therapy within 3 weeks prior to treatment
* Pregnant
* Lactating
* Presence of human anti-mouse antibody (HAMA) reactivity in patients with prior exposure to murine antibodies or proteins
* Serious nonmalignant disease or infection, which, in the opinion of the investigator, would compromise other protocol objectives
* Another primary malignancy (other than squamous cell and basal cell carcinoma of the skin, in situ carcinoma of the cervix, or treated prostate cancer with stable prostate specific antigen levels) for which the patients has not been disease-free for at least 3 years
* Major surgery, other than diagnostic surgery, within 4 weeks
* Patients with pleural effusion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-09; Primary Completion 2010-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Knox, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bexxar: Phase 2 study in patients with relapsed/refractory DLCL who were not candidates for transplantation. Bexxar was dosed as per the FDA approved regimen for other indications.
Period: Overall Study
Arm/Group | Bexxar
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bexxar
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate
Description: Clinical response rate for all participants, reported as the sum of the numbers of patients achieving complete response (CR, complete disappearance of all lesions); functional CR (fCR, minimal residual disease but clear of disease by positron emission tomography (PET)-scan); or partial response (PR, ≥ decrease in size of lesions and negative for active disease by PET-scan). Progressive disease (PD, advancing cancer) or stable disease (not CR, fCR, or PD) not included as Clinical Response.
Time Frame: 6 years
Measure: Number; unit: participants
Groups:
- Bexxar: Phase 2 study in patients with relapsed/refractory DLCL who were not candidates for transplantation. Bexxar was dosed as per the FDA-approved regimen for other indications.
Arm/Group | Bexxar
Number analyzed (Participants) | 9
participants
  Clinical Response | 2
  Complete Response (CR) | 0
  Functional CR | 1
  PR | 1
  SD | 6
  PD | 1

2. Secondary Outcome: Time to Progression (TTP)
Description: Time of disease progression reported as the number of subjects experiencing disease progression at the time point of progression.
Time Frame: 1.5 months; 3 months; 6 months; or Not Progressed
Population: 1 of the 9 study participants was lost-to-follow-up, and did not contribute data to this outcome.
Measure: Number; unit: participants
Arm/Group | Bexxar
Number analyzed (Participants) | 8
participants
  1.5 months | 1
  3 months | 2
  6 months | 2
  Not Progressed | 3

3. Secondary Outcome: Overall Survival (OS) Rate
Description: Overall survival reported as the percentage of participants (less lost-to-follow-up) surviving at 6 years.
Time Frame: 6 years
Population: 1 of the 9 study participants was lost-to-follow-up, and did not contribute data to this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Bexxar
Number analyzed (Participants) | 8
percentage of participants | 37.5

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Bexxar + Tylenol + Benadryl + SSKI: Bexxar is a radioimmunotherapeutic drug, an antibody that specifically attaches to the CD20 antigen, which is present on the surfaces of B cells and B cell lymphoma cells. Bexxar is patient specific: 75 cGy whole body patients with platelet count of 150,000/mm³ and 65 cGy for patients with platelet count less than 150,000/mm³, IV
Arm/Group | Bexxar + Tylenol + Benadryl + SSKI
Serious Adverse Events (participants affected / at risk) | 9/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexxar + Tylenol + Benadryl + SSKI (N=9)
Neutropenia (Blood and lymphatic system disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (1)
Stricture (Gastrointestinal disorders) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (1)
Thromnocytopenia (Blood and lymphatic system disorders) | 1 (1)
Stenosis (including anastomotic GI- Blilary tree) (Gastrointestinal disorders) | 1 (1)
Anemia-tachycardia (Blood and lymphatic system disorders) | 1 (1)
hypotension (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytoperia (Blood and lymphatic system disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexxar + Tylenol + Benadryl + SSKI (N=9)
Anemia (Blood and lymphatic system disorders) | 9 (9)
Back pains (Musculoskeletal and connective tissue disorders) | 5 (5)
Blurred visiom (Eye disorders) | 1 (1)
Burning Throat after SSKI (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Diarrehea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 9 (9)
Fatigue secondary to dexamethasone (General disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Foot Numbness (Nervous system disorders) | 1 (1)
High Neutrophil count (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) — (High BP ~155/103)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left side is sore (General disorders) | 1 (1)
Leg Swelling during the day (General disorders) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2)
Leukocytoperia (Blood and lymphatic system disorders) | 9 (9)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Loose Stools (Gastrointestinal disorders) | 1 (1)
Loss of balance (Ear and labyrinth disorders) | 2 (2)
Low Potassium (Metabolism and nutrition disorders) | 1 (1)
Memory Loss (Nervous system disorders) | 1 (1)
Mild headaches (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Neck Irritated (Skin and subcutaneous tissue disorders) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutroperia (Blood and lymphatic system disorders) | 7 (7)
Numbness (Musculoskeletal and connective tissue disorders) | 4 (4) — in legs and arms
Pain (General disorders) | 3 (3) — within body
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Renal insufficiency (Investigations) | 1 (1) — Increase Creatinine
Swelling (General disorders) | 4 (4) — within the body (arms, legs, groin,etc)
Throbbing Intermittent (Musculoskeletal and connective tissue disorders) | 4 (4) — within the groin area
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (9)
Upset Stomach (Gastrointestinal disorders) | 1 (1)
Skin Cancers (Skin and subcutaneous tissue disorders) | 1 (1) — sideburns, arms, all removed
Small cold (Gastrointestinal disorders) | 1 (1) — (runny nose, tired)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No